CLINICAL TRIAL: NCT03988192
Title: Volatile Organic Compounds in Exhaled Air and Sweat of Patients Treated by Immunotherapy for Lung Cancer: Research on Biomarkers for Early Therapeutic Response
Acronym: Immuno-VOC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Evolution of the treatment procedures so that their is no more benefits for patients
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018042
Record Dates: First submitted 2018-10-05; First posted 2019-06-17 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Lung Cancer, Non-small Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VOC analysis (Experimental): VOC analysis in exhaled air and sweat in patients treated by immunotherapy for lung cancer.
  Interventions: Device: VOC analysis

INTERVENTIONS:
Device: VOC analysis — VOC analysis in exhaled air with e-noses and mass spectrometry.

SUMMARY:
The study of volatile organic compounds (VOC) detected in exhaled air or in sweat, is an innovative research area for respiratory diseases. The volatolomic analysis can be done either by the technique of the mass spectrometry which allows the identification of each VOC in the exhaled air or by the technique of electronic nose, simpler and faster, which provides an idea of the general profile of the VOC without identifying them. The VOC have shown their interest in some situations, such as diagnostic or prognostic tool in patients followed for thoracic tumorous pathology or bronchial or pulmonary vascular diseases.

Immunotherapy is a new therapeutic approach used in non small cell lung cancer in a late stage.

VOC analysis could allow to identify biomarkers of early response to immunotherapy. The study of VOC could help in the optimisation of immunotherapy prescription in lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* patient aged > 18 years old
* patient with metastatic non-small cell lung cancer with marketing authorisation criteria for immunotherapy
* preserved overall condition (Performans Status 1)
* signed informed consent
* patient with healthcare insurance

Non Inclusion Criteria:

* patient with oxygen therapy or invasive ventilation
* patient unable to perform a slow vital capacity
* systemic corticosteroid therapy more than 10 mg per day of prednisone equivalent
* previous treatment with immunotherapy
* dermatological therapy interfering with sweat collection (psoriasis, irritant dermatitis, for instance)
* Patient deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Profiles of Volatil Organic Compound (VOC) in exhaled air | 1 day
  Comparison of variation of Volatil Organic Compound (VOC) profiles in exhaled air of patients before and during immunotherapy
Variation of Volatil Organic Compound (VOC) in exhaled air | change from baseline profiles at week 9, week 18 and week 27 post-baseline
  Correlation of variation with response to immunotherapy at week 9, 18 and 27 (according to RECIST criteria)

SECONDARY OUTCOMES:
Profiles of Volatil Organic Compound (VOC) in sweat | 1 day
  Comparison of variation of Volatil Organic Compound (VOC) profiles in sweat of patients before and during immunotherapy
Variation of Volatil Organic Compound (VOC) in sweat | change from baseline profiles at week 9, week 18 and week 27 post-baseline
  Correlation of variation with response to immunotherapy at week 9, 18 and 27 (according to RECIST criteria)
Volatil Organic Compound (VOC) profile and radiological response | change from baseline profiles at week 9, week 18 and week 27 post-baseline
  Correlation between Volatil Organic Compound (VOC) profile before treatment and radiological response at 9, 18 and 27 weeks (defined by RECIST criteria)
Volatil Organic Compound (VOC) profile and drug toxicity | change from baseline profiles at week 9, week 18 and week 27 post-baseline
  Correlation between variation of Volatil Organic Compound (VOC) profiles and apparition of drug toxicity at 9, 18 and 27 weeks
Comparison of performance from Volatil Organic Compound (VOC) from exhaled air versus sweat | 1 day
  Comparison of performance of Volatil Organic Compound (VOC) from exhaled air versus Volatil Organic Compound (VOC) from sweat
Comparison of performance of mass spectrometry versus electronic noses | 1 day
  Comparison of performance of Volatil Organic Compound (VOC) from mass spectrometry versus Volatil Organic Compound (VOC) from electronic noses

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Devillier, Principal Investigator — Pneumology department
Locations (1):
- Hôpital Foch, Suresnes, France